CLINICAL TRIAL: NCT00484874
Title: A Phase I/II Study of I-131 Tositumomab in Patients With Relapsed/Refractory Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of I-131 Tositumomab in Patients With Relapsed/Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0703; NA_00005743 (Other: JHM IRB)
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin's lymphoma; Radioimmunotherapy; Bexxar; I-131 Tositumomab; Safety; Efficacy; Nuclear Medicine; Monoclonal antibody; Radiolabeled
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- A Single Dose of I-131 Tositumomab (Experimental): I-131 Tositumomab therapeutic regimen given to patients with relapsed/refractory Hodgkin's lymphoma who have or have not undergone transplant.
  Interventions: Drug: I-131 Tositumomab therapeutic regimen

INTERVENTIONS:
Drug: I-131 Tositumomab therapeutic regimen — Tositumomab and I-131 tositumomab are given intravenously. A test dose is given followed by a larger treatment dose.
  Other Names: Brand name: Bexxar

SUMMARY:
The purpose of this study is to find the highest safe dose of Iodine-131 Tositumomab (Bexxar®) that can be given to patients who have relapsed/refractory Hodgkin's lymphoma, what side effects these patients get when they take Bexxar® and if Bexxar® is effective in treating relapsed/refractory Hodgkin's lymphoma. Bexxar® works by delivering doses of radiation to cancer cells.

DETAILED DESCRIPTION:
One third of patients with Hodgkin's lymphoma (HL) do not respond to or have their disease come back after their first therapy. These patients often then receive high-dose chemotherapy and blood or marrow transplant. Despite high response rates after transplant, a significant number, 26-65%, of these patients have their disease come back again. After transplant, therapy options are limited and alternative therapies for patients with HL who have relapsed post-transplant or who are ineligible for transplant are needed. Based on recent studies about how HL develops and good results of patient studies evaluating the use of the unlabeled anti-CD20 antibody Rituximab in HL, we think that radioimmunotherapy (RIT) with I-131 Tositumomab(Bexxar®) will be an effective alternative therapy in patients with relapsed/refractory HL who are post or ineligible for transplant.

The rationale for the use of RIT in cancer is that radiolabeled monoclonal antibodies will specifically target and irradiate tumor cells but not normal tissues. The specific tumor targeting of RIT theoretically allows higher doses of radiation to be delivered to tumor as compared to external beam radiation because the effects of the radiation on normal tissues is less with RIT. Iodine-131 Tositumomab (Bexxar®) was approved by the FDA for another type of lymphoma in 2003. The antibody (Tositumomab) recognizes and attaches to a protein on lymphoma cells and can kill these cells. The radioisotope (I-131) can help the antibody kill cells better.

Iodine-131 Tositumomab (Bexxar®) is given through a vein in the arm. Iodine-131 Tositumomab (Bexxar®) is given in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Hodgkin's lymphoma that is relapsed or refractory and the patient has previously had a transplant or is ineligible for transplant
* All stages and histologic subtypes of Hodgkin's lymphoma
* Malignant cells may be CD20+ or CD20-
* May have previously had either a non-myeloablative or myeloablative allogeneic or autologous stem cell transplant
* If prior history of greater than 1 transplant, eligible if other entry criteria are met
* No upper limit on the amount of prior chemotherapy
* Must be at least 4 weeks out from their most recent chemotherapy or radiation therapy, 6 weeks if the last regimen included BCNU, or mitomycin
* Age 18 or greater
* Karnofsky performance status ≥ 60
* Organ and marrow function within 4 weeks of registration on the protocol as defined below:
* Leukocytes >2,000/mm3
* Absolute neutrophil count >1,000/ mm3
* Platelets >75,000/ mm3
* Hemoglobin >7 g/dL
* Creatinine <2.5 mg/dL
* Less than 25% bone marrow involvement with Hodgkin's lymphoma within 4 weeks of registration on the protocol
* If female, not pregnant or breast feeding
* Ability to understand and the willingness to sign a written informed consent document
* At least one measurable target lesion, measuring 1.5 cm in at least one dimension by standard CT imaging which is FDG -avid on PET/CT.
* 2-year expected survival from other diseases

Exclusion Criteria:

* Receiving any other investigational agents at the same time
* Hypocellular bone marrow (less than or equal to 10% cellularity) or marked decrease in any one (or more) hematopoietic precursor within 4 weeks of registration on the protocol
* Inability to follow basic radiation safety precautions
* Active infections requiring intravenous antibiotics until after resolution of the infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2014-01 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wahl, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A Single Dose of I-131 Tositumomab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | A Single Dose of I-131 Tositumomab
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 36 [20 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Post-transplant [Count of Participants; unit: Participants] — Previously received blood or marrow transplant.
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: Non-myeloablative Maximum Tolerated Dose of I-131 Tositumomab That Can be Given to Patients With Relapsed/Refractory Hodgkin's Lymphoma.
Time Frame: 2 years
Measure: Number; unit: cGy
Groups:
- A Single Dose of I-131 Tositumomab: Non-myeloablative maximum tolerated dose of I-131 Tositumomab that can be given to patients with relapsed/refractory Hodgkin's lymphoma.
  I-131 Tositumomab therapeutic regimen: Tositumomab and I-131 tositumomab are given intravenously. A test dose is given followed by a larger treatment dose.
Arm/Group | A Single Dose of I-131 Tositumomab
Number analyzed (Participants) | 12
cGy | 79

2. Primary Outcome: Overall and Complete Response Rates
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CTI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 12 weeks post therapy
Measure: Number; unit: percentage of participants
Groups:
- A Single Dose of I-131 Tositumomab: A single therapeutic dosage of 131I-tositumomab.
  I-131 Tositumomab therapeutic regimen: Tositumomab and I-131 tositumomab are given intravenously. A test dose is given followed by a larger treatment dose.
Arm/Group | A Single Dose of I-131 Tositumomab
Number analyzed (Participants) | 12
percentage of participants
  ORR | 25
  CRR | 25

3. Secondary Outcome: Median Time to Progression Following I-131 Tositumomab Therapy.
Time Frame: From time measurement criteria are met for response until first date that recurrent or progressive disease is objectively documented, assessed up to 5 years.
Measure: Median (Standard Deviation); unit: weeks
Groups:
- A Single Therapeutic Dosage of 131I-tositumomab: A single therapeutic dosage of 131I-tositumomab in patients who have undergone transplant.
  I-131 Tositumomab therapeutic regimen: Tositumomab and I-131 tositumomab are given intravenously. A test dose is given followed by a larger treatment dose.
Arm/Group | A Single Therapeutic Dosage of 131I-tositumomab
Number analyzed (Participants) | 12
weeks | 12 (3.3)

4. Secondary Outcome: Frequency of Visualization of Hodgkin's Lymphoma With I-131 Tositumomab Imaging and Tumor Radiation Absorbed Dose
Description: Percentage of participants with visualized I-131 uptake.
Time Frame: up to 1 week post-intervention
Measure: Number; unit: Percentage of patients with I-131 uptake
Groups:
- Treatment: A single therapeutic dosage of 131I-tositumomab.
  I-131 Tositumomab therapeutic regimen: Tositumomab and I-131 tositumomab are given intravenously. A test dose is given followed by a larger treatment dose.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Percentage of patients with I-131 uptake | 100

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 2 years following the administration of I-131 Tositumomab.
Arm/Group | A Single Dose of I-131 Tositumomab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Single Dose of I-131 Tositumomab (N=12)
Hemoglobin Decreased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 4
Platelet Count Decreased (Investigations) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Single Dose of I-131 Tositumomab (N=12)
Hemoglobin Decreased (Investigations) | 6
Anemia (Blood and lymphatic system disorders) | 1
Platelet Count Decreased (Investigations) | 6
Fatigue (General disorders) | 5
Lungm aero-digestive (Infections and infestations) | 1
Hypothyroidism (Endocrine disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Fever (General disorders) | 1
Chills (General disorders) | 1
Cold Intolerance (General disorders) | 1
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No